CLINICAL TRIAL: NCT06609785
Title: The Relationship Between Exercise-drived Exosomes and Diabetes Mellitus.
Brief Title: Differential Regulation of miRNA and Protein in Human Plasma Extracellular Vesicles by Different Types of Exercise.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xiaofeng Zheng, principal investigator, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022629
Record Dates: First submitted 2024-09-19; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Diabetes; Exercise; Lifestyle Intervention
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise training group (Experimental): All volunteers had a standardized breakfast, and all tests started at 9:00 a.m. The volunteers successively completed both high intensity interval training (HIIT) and continuous aerobic training (CAT) under the supervision of a professional coach, and the interval between each type of exercise was 7 days. Each training session was initiated with a brief 2-minute standardized warm-up, followed by 20 minutes of cycling consisting of periods of 2 minutes at 80-95% maximal heart rate (HRmax) separated by 2 minutes of active recovery for the HIIT group or 20 minutes of cycling at 60-80% of HRmax for the CAT group. A real-time heart rate monitoring system was continuously used during each training session.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The volunteers successively completed both high intensity interval training (HIIT)and continuous aerobic training (CAT) under the supervision of a professional coach, and the interval between each type of exercise was 7 days. Each training session was initiated with a brief 2-minute standardized warm-up, followed by 20 minutes of cycling consisting of periods of 2 minutes at 80-95% maximal heart rate (HRmax) separated by 2 minutes of active recovery for the HIIT group or 20 minutes of cycling at 60-80% of HRmax for the CAT group.

SUMMARY:
Aims/hypothesis: Both continuous aerobic training (CAT) and high intensity interval training (HIIT) are recommended to promote health and prevent diseases. Exercise-induced circulating extracellular vesicles (EX-EVs) have been suggested to play essential roles in mediating organ crosstalk, but corresponding molecular mechanisms remain largely unexplored. We aimed to assess and compare the systemic effects of CAT and HIIT via multi-omics integration analysis of EX-EVs.

Methods: Five healthy male volunteers were assigned to HIIT (20 minutes of cycling with periods of 2 minutes at 80-95% HRmax separated by 2 minutes of active recovery) and CAT (20 minutes of cycling at 60-80% of HRmax), with a 7-day interval between sessions. Plasma EVs were collected at rest or immediately after each training section, prior to proteomics and miRNA profile analysis.

DETAILED DESCRIPTION:
Before the formal experiment, the volunteers were undergoing a thorough physical examination and proper training to ensure that they were able to complete the experiment. The participants refrained from exercise 24 hours prior to the test to ensure the integrity and accuracy of the results. All volunteers had a standardized breakfast, and all tests started at 9:00 a.m. The volunteers successively completed both HIIT and CAT under the supervision of a professional coach, and the interval between each type of exercise was 7 days. Each training session was initiated with a brief 2-minute standardized warm-up, followed by 20 minutes of cycling consisting of periods of 2 minutes at 80-95% maximal heart rate (HRmax) separated by 2 minutes of active recovery for the HIIT group or 20 minutes of cycling at 60-80% of HRmax for the CAT group. A real-time heart rate monitoring system was continuously used during each training session. The participants were instructed to continue their regular physical activities and eating habits throughout the intervention period. Blood samples were collected at rest or immediately after each training session for further analysis.

ELIGIBILITY:
Inclusion Criteria:

18-65 years of age Body mass index (BMI) values between 18-28 kg/m2 More than 3 h of physical activity per week Acknowledgment of informed consent.

-

Exclusion Criteria:

Smokers Body weight change >5 kg in 6 months Unsuitable for physical training (heart disease, respiratory disorders or any conditions that could be aggravated by exercise) Currently taking medication or having a history of medication such as steroids, beta-blockers or anticoagulants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
miRNA and proteins in human plasma-derived extracellular vesicles | From enrollment to the end of intervention at 2 weeks
  Measuring miRNA and proteins in human plasma-derived extracellular vesicles through high-throughput sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Per-Olof Berggren, Principal Investigator — Department of Molecular Medicine and Surgery, Karolinska Institutet, SE-17177 Stockholm, Sweden
Locations (1):
- Department of Endocrinology and Metabolism, Research Center for Islet Transplantation, West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Time Frame: Beginning 1 year and ending 3 years after publication
Access Criteria: Any researchers who has undergone an approval process will be able to access the IPD and supporting information, Applicants are required to submit a data use application via the following email( yrou2001@163.com ),including the research plan and other relevant documents. Once approved , the applicant will receive the data via a secure file transfer method.